CLINICAL TRIAL: NCT06352190
Title: An Open-Label, Single-Center, Single-Dose, Phase I Study to Assess the Mass Balance of [14C] SY-5007 in Healthy Male Subjects in China
Brief Title: A Study to Evaluate the Mass Balance of [14C] SY-5007 in Healthy Adult Male Subjects in China
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shouyao Holdings (Beijing) Co. LTD (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SY-5007-I-04
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2023-12

CONDITIONS: Healthy Subjects
Keywords: [14C] SY-5007; Mass Balance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SY-5007 (Experimental): Single oral dose of 160 mg SY-5007 suspension (containing approximately 120 μCi [14C] SY-5007)
  Interventions: Drug: [14C] SY-5007

INTERVENTIONS:
Drug: [14C] SY-5007 — Carbon-14 labeled SY-5007

SUMMARY:
This is a single-center, open-label, non-randomized, single dose study in healthy male subjects designed to assess mass balance recovery, metabolite profile and metabolite identification of radio-labeled SY-5007 administered orally.

DETAILED DESCRIPTION:
The trial will consist of two parts:

Pilot Study:

Two eligible adult male subjects will be enrolled and admitted to the clinical trial center after passing the inclusion criteria review. They will undergo training on medication administration, urine and feces collection, etc., to ensure compliance with the protocol and standard operating procedures (SOP). Subjects will fast before medication administration and provide urine and feces samples at specified intervals after dosing. Blood samples will also be collected at specified time points.

Formal Study:

Four to six male subjects will be enrolled, receiving a single dose of SY-5007 160 mg orally containinig roughly 120 µCi [14C] SY-5007. Blood, urine and feces samples will be collected at specified time points.

Safety monitoring (12-lead ECG, vital signs, blood chemistry and haematology) and adverse events will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be enrolled in this study:

1. Fully informed, able to communicate effectively with researchers, agree to abide by the protocol and trial management regulations, and voluntarily sign the written Informed Consent Form (ICF);
2. Healthy adult males aged 18 to 50 years at the time of signing the ICF, with no plans for reproduction or sperm donation within the past 2 years;
3. Weight ≥ 50 kg and body mass index (BMI) between 18 and 26 kg/m2;
4. Subjects of reproductive capability agree to employ effective contraceptive measures with their sexual partners during the study period and for 2 years following the end of the study.

Exclusion Criteria:

Subjects meeting any of the following criteria are ineligible for participation in this study:

1. History of allergies (such as allergies to two or more drugs, foods, or pollen, or individuals prone to skin hives or allergic reactions).
2. Positive for hepatitis B surface antigen, hepatitis C virus antibodies, human immunodeficiency virus antibodies, or positive for syphilis treponemal and non-treponemal antibodies during screening.
3. Abnormal clinically significant vital signs, physical examinations, laboratory tests, or electrocardiograms at screening.
4. Gastrointestinal, hepatic, or renal diseases that may affect drug pharmacokinetics as assessed by the investigator at screening.
5. History of drug abuse or illicit drug use within 12 months prior to the first dose administration, or positive urine drug screening test during screening.
6. Underwent major surgery within 6 months prior to the first dose administration, or planned to undergo surgery during the trial period.
7. History of any clinically significant illness within 3 months prior to the first dose administration or conditions deemed by the investigator to potentially affect trial outcomes, including but not limited to cardiovascular, endocrine, nervous, respiratory, digestive, urinary, hematologic, immune, or psychiatric disorders.
8. Average daily smoking of more than 5 cigarettes within 3 months prior to the first dose administration, or unwillingness to discontinue use of any tobacco products during the trial.
9. Regular alcohol consumption within 3 months prior to the first dose administration [defined as consuming more than 14 units of alcohol per week (1 unit = 360mL of 5% alcohol beer or 45mL of 40% alcohol liquor or 150mL of 12% alcohol wine)], or inability to abstain from alcohol during the trial, or positive alcohol breath test during screening.
10. History of blood donation or significant blood loss (≥ 300mL) within 3 months prior to the first dose administration, or use of blood products or blood transfusion within 1 month prior to the first dose administration.
11. Participation in other drug or medical device clinical trials within 3 months prior to the first dose administration (excluding screen failures), or prior use of the investigational drug.
12. Vaccination within 1 month prior to the first dose administration.
13. Use of any prescription drugs, over-the-counter drugs, supplements, or herbal remedies within 2 weeks prior to the first dose administration (if the half-life [t1/2] of the drug can be confirmed, a washout period of 5 times of t1/2 is required).
14. Habitual consumption of more than 8 cups (1 cup = 250mL) of tea, coffee, or caffeinated beverages and unable to abstain from consumption within 48 hours prior to the first dose administration and during the trial.
15. Special dietary requirements or difficulty swallowing.
16. Habitual constipation or previous difficulty with bowel movements.
17. Difficulty with blood collection, history of fainting with needles, or intolerance to venipuncture.
18. Engagement in occupations requiring prolonged exposure to radioactive conditions; or significant exposure to radiation within 1 year prior to the trial (e.g., 2 chest/abdominal CT scans, or 3 other types of X-ray examinations).
19. History of definite neurological or psychiatric disorders, including dementia or seizures diagnosed for any reason.
20. Other conditions deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Total radioactivity in plasma PK: Cmax | At pre-dose and up to 2 weeks post-dose
  Highest radioactivity observed plasma concentration
Total radioactivity in plasma PK: Tmax | At pre-dose and up to 2 weeks post-dose
  Time to reach the Cmax
Total radioactivity in plasma PK: AUC0-t | At pre-dose and up to 2 weeks post-dose
  Defined as area under the single-dose plasma concentration-time curve from Hour 0 to the last quantifiable measurable plasma concentration
Total radioactivity in plasma PK: t½ | At pre-dose and up to 2 weeks post-dose
  Defined as apparent plasma terminal phase disposition half-life
Total radioactivity in plasma PK: CL/F | At pre-dose and up to 2 weeks post-dose
  Defined as apparent total body clearance
Whole blood to plasma total radioactivity ratio | At pre-dose and up to 2 weeks post-dose
  To evaluate the extent of distribution of total radioactivity into blood cells
Cumulative total radioactivity in urine and faeces | At pre-dose and up to 2 weeks post-dose
  Mass balance recovery of total radioactivity in all (urine, faeces) amount excreted (Ae) expressed as a percentage of the administered dose (%Ae)
Metabolic profiling in plasma, urinary and fecal excretion | At pre-dose and up to 2 weeks post-dose
  To characterize the metabolic profile and identify circulating and excreted metabolites of SY-5007 using liquid chromatography with mass spectral detection.

SECONDARY OUTCOMES:
Cmax of SY-5007 and its metabolites | At pre-dose and up to 2 weeks post-dose
  Defined as maximum observed plasma concentration
Tmax of SY-5007 and its metabolites | At pre-dose and up to 2 weeks post-dose
  Defined as time to maximum plasma concentration
AUC0-t of SY-5007 and its metabolites | At pre-dose and up to 2 weeks post-dose
  Defined as area under the single-dose plasma concentration-time curve from Hour 0 to the last quantifiable measurable plasma concentration
t½ of SY-5007 and its metabolites | At pre-dose and up to 2 weeks post-dose
  Defined as apparent plasma terminal phase disposition half-life
CL/F of SY-5007 and its metabolites | At pre-dose and up to 2 weeks post-dose
  Defined as apparent total body clearance
Incidence of adverse events | At pre-dose and up to 2 weeks post-dose
  To evaluate the safety of a single oral dose of 160 mg of SY-5007

CONTACTS AND LOCATIONS:
Overall Officials: Yinghui Sun, PhD, Study Director — Shouyao Holdings (Beijing) Co. LTD
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, China